CLINICAL TRIAL: NCT03127241
Title: USEFUL: User-centred Assistive SystEm for Arm Functions in neUromuscuLar Subjects
Brief Title: User-centred Assistive System for Arm Functions in Neuromuscular Subjects
Acronym: USEFUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Politecnico di Milano (Other)
Collaborators: IRCCS Eugenio Medea (Other); Villa Beretta Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Alessandra Pedrocchi, Professor, Politecnico di Milano
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: GUP 15021
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Dystrophy, Becker; Muscular Dystrophy, Limb-Girdle Type 2
Keywords: Assistive devices; Randomized controlled trial (RCT); Upper limbs; Robotic devices
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne; Limb-girdle muscular dystrophy type 2A | interventions — Self-Help Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Armon Ayura (Active Comparator): Upper limb assistive device with active solutions for gravity compensation. Intervention: The upper limb exoskeleton is worn by the patient on the preferred arm, and it is used during daily life activities to support arm movements, particularly getting rid of gravity arm weight.
  Interventions: Device: Assistive device (Armon Ayura) test
- Jaeco Wrex (Active Comparator): Upper limb assistive device with passive solutions for gravity compensation. Intervention: The upper limb exoskeleton is worn by the patient on the preferred arm, and it is used during daily life activities to support arm movements, particularly getting rid of gravity arm weight.
  Interventions: Device: Assistive device (Jaeco Wrex) test

INTERVENTIONS:
Device: Assistive device (Armon Ayura) test — Short Training (T0-T1) - each subject will undergo a 3-day training at the clinical center during which technicians, along with a physiotherapist will adjust and customize the device and explain possible independent use at home.
  Domestic use (T1-T2) - Subjects will use the device during their daily life activities for two weeks at home. They will perform task-oriented movements (e.g. reaching a mouse and objects on a table, moving back to the wheelchair, drinking), free movements, playful activities (e.g. playing chess, leafing through a book), and self-care activities, accordingly to subject's residual capability, for a minimum period of 5 hours/day. They will keep a structured diary where all the problems, achievements and comments will be reported.
  Arms: Armon Ayura
Device: Assistive device (Jaeco Wrex) test — Short Training (T0-T1) - each subject will undergo a 3-day training at the clinical center during which technicians, along with a physiotherapist will adjust and customize the device and explain possible independent use at home.
  Domestic use (T1-T2) - Subjects will use the device during their daily life activities for two weeks at home. They will perform task-oriented movements (e.g. reaching a mouse and objects on a table, moving back to the wheelchair, drinking), free movements, playful activities (e.g. playing chess, leafing through a book), and self-care activities, accordingly to subject's residual capability, for a minimum period of 5 hours/day. They will keep a structured diary where all the problems, achievements and comments will be reported.
  Arms: Jaeco Wrex

SUMMARY:
Restore a lost function is a special experience for people affected by neuromuscular evolutive diseases. "From the patient's point of view improvement is measured by regaining lost abilities,-by being able to do something -anything-today I couldn't do yesterday ". Upper limb pain, stiffness and activity limitations have a crucial role in reducing patients' autonomy and worsening quality of life.

Real users' needs have been identified thought several workshops, and even if the commercial products might assure a benefit to some users and meet most of their requirements, so far a validation of the use of such devices by people with neuromuscular disease is missing.

We aim at field-testing the improvement in arm functions provided by the use of some commercial devices and assessing their impact to users' quality of life and independence. This step is essential to assure a widespread accessibility to these devices for most of the potential users, possibly providing health providers with direction and guidance towards Health Technology Assessment.

Clinical Trial design - The study proposes on-field validation of JAECO WREX, passive antigravity exoskeleton; and Armon Ayura, motorized arm exoskeleton for gravity compensation in a randomized controlled trial with crossover design. The clinical study will is multi-centric, involving both MEDEA and VALDUCE, and received the Ethical Committee approval.

ELIGIBILITY:
Inclusion criteria

* signed informed consent (we will expose the family the aims of our study and carefully describe the need of compliance with them)
* diagnosis of muscular dystrophy (genetic, histological and biochemical if necessary),specifically with Duchenne, Becker and Limb Girdle type 2 muscular dystrophy. No muscle biopsy will be performed, except in case there is a diagnostic need.
* being wheelchair bound
* having a scoring at the MRC scale for upper limb at the deltoid, biceps, triceps brachii muscles ranging from 2 to 4.

Exclusion criteria

* presence of additional diseases (for example: family history of mental retardation, epilepsy, cerebral palsy)
* behavioral and psychiatric disturbances (emotional problems, depression)
* absence of compliance to the study of the family and the caregivers

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Performance of the Upper Limb (PUL) scale | T0 (baseline); T1 (after 3-days short training with device 1); T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  The PUL includes 22 items with an entry item to define the starting functional level, and 21 items subdivided into shoulder level (4 items), middle level (9 items) and distal level (8 items) dimension. For weaker patients a low score on the entry item means high level items do not need to be performed. Scoring options vary across the scale between 0-1 to 0-6 according to performance. Each dimension can be scored separately with a maximum score of 16 for the shoulder level, 34 for the middle level, and 24 for the distal level . A total score can be achieved by adding the three level scores (max total score 74).

SECONDARY OUTCOMES:
Motor Function Measures scale (MFM) | T0 (baseline); T1 (after 3-days short training with device 1); T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  MFM is a quantitative scale that makes it possible to measure the functional motor abilities of a person affected by a neuromuscular disease.
Brooke scale | T0 (baseline); T1 (after 3-days short training with device 1); T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  The Brooke scale was designed to assess the upper extremity function. The grades of the Brooke scale range from 1 to 6; 1 means that the subject can elevate their arms full range to the head with the arms straight; while 2 means that the shoulder strength is insufficient to elevate their arms and the subject needs to flex the elbow to elevate the arms; in grades 3 and 4, the subject is unable to elevate the shoulders but can raise hands to the mouth with or without weight respectively; grade 5 refers to the subject being unable to raise hands to the mouth and only some hand movement exists, while grade 6 refers to no useful function of hands.
ABILHAND | T0 (baseline); T1 (after 3-days short training with device 1); T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  a measure of manual ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved
PedsQL | T0 (baseline); T2 (after 2-weeks home use of device 1 - primary assessment point); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  Neuromuscular module: composed of 25 items comprising 3 dimensions, i.e. about my neuromuscular disease (1-17); communication (1-3); and about our faily resources (1-5) Multidimensional Fatigue module: composed of 18 items comprising 3 dimensions, i.e. general fatigue (1-6); sleep/rest fatigue (1-6); and cognitive fatigue (1-6).
PROMIS FATIGUE Short Form | T0 (baseline); T2 (after 2-weeks home use of device 1 - primary assessment point); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  The PROMIS Fatigue instruments evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The Fatigue short form is universal rather than disease-specific. It assesses fatigue over the past seven days.
Personal Adjustment and Role Skills Scale (PARS) III | T0 (baseline); T2 (after 2-weeks home use of device 1 - primary assessment point); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  PARS III to assesses the psychosocial adjustment of children with chronic physical illnesses and no mental impairment. The PARS III consists of 28 items that measure psychosocial functioning in six areas: peer relations, dependency, hostility, productivity, anxiety-depression, and withdrawal.
Technology Acceptance Model (TAM) | T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  Technology Acceptance Model (TAM) provides a valid and reliable measure that predicts the acceptance or adoption of new technologies by end-users. TAM predicts acceptance based on the end-user's perceived usefulness (6 items) and perceived ease of use (6 items) of the technology for a specific purpose.
System Usability Scale (SUS) | T2 (after 2-weeks home use of device 1 - primary assessment point); T3 (after 3-days short training with device 2); T4 (after 2-weeks home use of device 2 - secondary assessment point)
  the system usability scale (SUS) is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. Measurements of usability have several different aspects: effectiveness (can users successfully achieve their objectives); efficiency (how much effort and resource is expended in achieving those objectives); and satisfaction (was the experience satisfactory).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Pedrocchi, Prof, Principal Investigator — Politecnico di Milano
Locations (2):
- Italy (2):
  - IRCCS E. Medea - La Nostra Famiglia, Bosisio Parini, LC
  - Villa Beretta, Costa Masnaga, LC

REFERENCES:
- [Background] Magri F, Nigro V, Angelini C, Mongini T, Mora M, Moroni I, Toscano A, D'angelo MG, Tomelleri G, Siciliano G, Ricci G, Bruno C, Corti S, Musumeci O, Tasca G, Ricci E, Monforte M, Sciacco M, Fiorillo C, Gandossini S, Minetti C, Morandi L, Savarese M, Fruscio GD, Semplicini C, Pegoraro E, Govoni A, Brusa R, Del Bo R, Ronchi D, Moggio M, Bresolin N, Comi GP. The italian limb girdle muscular dystrophy registry: Relative frequency, clinical features, and differential diagnosis. Muscle Nerve. 2017 Jan;55(1):55-68. doi: 10.1002/mus.25192. Epub 2016 Oct 28. PMID 27184587
- [Background] Ricci G, Ruggiero L, Vercelli L, Sera F, Nikolic A, Govi M, Mele F, Daolio J, Angelini C, Antonini G, Berardinelli A, Bucci E, Cao M, D'Amico MC, D'Angelo G, Di Muzio A, Filosto M, Maggi L, Moggio M, Mongini T, Morandi L, Pegoraro E, Rodolico C, Santoro L, Siciliano G, Tomelleri G, Villa L, Tupler R. A novel clinical tool to classify facioscapulohumeral muscular dystrophy phenotypes. J Neurol. 2016 Jun;263(6):1204-14. doi: 10.1007/s00415-016-8123-2. Epub 2016 Apr 28. PMID 27126453
- [Background] Pane M, Mazzone ES, Fanelli L, De Sanctis R, Bianco F, Sivo S, D'Amico A, Messina S, Battini R, Scutifero M, Petillo R, Frosini S, Scalise R, Vita G, Bruno C, Pedemonte M, Mongini T, Pegoraro E, Brustia F, Gardani A, Berardinelli A, Lanzillotta V, Viggiano E, Cavallaro F, Sframeli M, Bello L, Barp A, Bonfiglio S, Rolle E, Colia G, Catteruccia M, Palermo C, D'Angelo G, Pini A, Iotti E, Gorni K, Baranello G, Morandi L, Bertini E, Politano L, Sormani M, Mercuri E. Reliability of the Performance of Upper Limb assessment in Duchenne muscular dystrophy. Neuromuscul Disord. 2014 Mar;24(3):201-6. doi: 10.1016/j.nmd.2013.11.014. Epub 2013 Dec 5. PMID 24440357
- [Background] McDonald CM, Meier T, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Spagnolo P, Buyse GM; DELOS Study Group. Idebenone reduces respiratory complications in patients with Duchenne muscular dystrophy. Neuromuscul Disord. 2016 Aug;26(8):473-80. doi: 10.1016/j.nmd.2016.05.008. Epub 2016 May 12. PMID 27238057
- [Background] Messina S, Vita GL, Sframeli M, Mondello S, Mazzone E, D'Amico A, Berardinelli A, La Rosa M, Bruno C, Distefano MG, Baranello G, Barcellona C, Scutifero M, Marcato S, Palmieri A, Politano L, Morandi L, Mongini T, Pegoraro E, D'Angelo MG, Pane M, Rodolico C, Minetti C, Bertini E, Vita G, Mercuri E. Health-related quality of life and functional changes in DMD: A 12-month longitudinal cohort study. Neuromuscul Disord. 2016 Mar;26(3):189-96. doi: 10.1016/j.nmd.2016.01.003. Epub 2016 Feb 2. PMID 26916554
- [Background] Pane M, Fanelli L, Mazzone ES, Olivieri G, D'Amico A, Messina S, Scutifero M, Battini R, Petillo R, Frosini S, Sivo S, Vita GL, Bruno C, Mongini T, Pegoraro E, De Sanctis R, Gardani A, Berardinelli A, Lanzillotta V, Carlesi A, Viggiano E, Cavallaro F, Sframeli M, Bello L, Barp A, Bianco F, Bonfiglio S, Rolle E, Palermo C, D'Angelo G, Pini A, Iotti E, Gorni K, Baranello G, Bertini E, Politano L, Sormani MP, Mercuri E. Benefits of glucocorticoids in non-ambulant boys/men with Duchenne muscular dystrophy: A multicentric longitudinal study using the Performance of Upper Limb test. Neuromuscul Disord. 2015 Oct;25(10):749-53. doi: 10.1016/j.nmd.2015.07.009. Epub 2015 Jul 17. PMID 26248957
- [Background] Magliano L, D'Angelo MG, Vita G, Pane M, D'Amico A, Balottin U, Angelini C, Battini R, Politano L, Patalano M, Sagliocchi A, Civati F, Brighina E, Vita GL, Messina S, Sframeli M, Lombardo ME, Scalise R, Colia G, Catteruccia M, Berardinelli A, Motta MC, Gaiani A, Semplicini C, Bello L, Astrea G, Zaccaro A, Scutifero M. Psychological and practical difficulties among parents and healthy siblings of children with Duchenne vs. Becker muscular dystrophy: an Italian comparative study. Acta Myol. 2014 Dec;33(3):136-43. PMID 25873782
- [Background] Buyse GM, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Mayer OH, Spagnolo P, Meier T, McDonald CM; DELOS Study Group. Treatment effect of idebenone on inspiratory function in patients with Duchenne muscular dystrophy. Pediatr Pulmonol. 2017 Apr;52(4):508-515. doi: 10.1002/ppul.23547. Epub 2016 Aug 29. PMID 27571420
- [Derived] Longatelli V, Antonietti A, Biffi E, Diella E, D'Angelo MG, Rossini M, Molteni F, Bocciolone M, Pedrocchi A, Gandolla M. User-centred assistive SystEm for arm Functions in neUromuscuLar subjects (USEFUL): a randomized controlled study. J Neuroeng Rehabil. 2021 Jan 6;18(1):4. doi: 10.1186/s12984-020-00794-z. PMID 33407580